CLINICAL TRIAL: NCT01780870
Title: Weight Loss Study-Mechanism Underlying the Improvement of Insulin Resistance in Response to Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Christos Mantzoros, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011P000293
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-05

CONDITIONS: Obesity; Weight Loss
Keywords: Overweight; Obesity; Obese; Weight loss
MeSH Terms: conditions — Obesity; Weight Loss; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Obese, otherwise healthy people who are not receiving any nutritional,surgical or behavioral therapy
- Weight loss group (Active Comparator): Full Meal replacement Protocol
  Interventions: Dietary Supplement: Weight loss group (Full meal replacement products)

INTERVENTIONS:
Dietary Supplement: Weight loss group (Full meal replacement products) — In the intervention arm of this non randomized, open label study to assess the effects of weight loss on insulin sensitivity and leptin tolerance subjects will use full meal replacement products (1280-1320kcal/day). Subjects will be on the full meal replacement products only, for the first 12 weeks, between 13 to 19 weeks they will be transitioned to regular food, from 19 weeks and going forward they will be on chronic maintenance phase
  Other Names: Full meal replacement products (1280-1320 kcal/day)
  Arms: Weight loss group

SUMMARY:
The main purpose of this study is to assess factors mediating the changes in insulin sensitivity and glucose tolerance before and after 10 lbs ± or 2% weight loss reduction as well as 2, 3, 6, 12, and 24 months after initiation of a low calorie diet.

The investigators will also study the following:

1. The impact of diet induced weight loss on hormones/adipokine levels
2. The impact of diet induced weight loss on leptin tolerance

ELIGIBILITY:
Inclusion Criteria for interventional group:

1. Adult men and women, age 18-50
2. English speaking
3. Body mass index (pre weight loss) ≥30 kg/m2 but <40 kg/m2
4. Willing to enroll in a low calorie full meal replacement weight loss program
5. Willing and able to take part in a multi year study involving visits

Inclusion Criteria for control group:

1. Adult men and women, age 18-50
2. English speaking
3. Body mass index (pre weight loss) ≥30 kg/m2 but <40 kg/m2
4. Willing and able to take part in a multi year study involving visits

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Mantzoros, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Weight Loss Group
Started | 0 | 5
Completed | 0 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to enrolling problems, no subjects were enrolled to the control group. All the subjects were enrolled to the weight loss group
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Weight Loss Group | Total
Number analyzed (Participants) | 0 | 5 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 5 | 5
  >=65 years |  | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 32.8 (3.1) | 32.8 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 5 | 5
  Male |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Will be the Leptin Levels at Baseline and 8 Weeks
Description: The secondary outcome was deleted, since it was finally not performed in the study due to problems in enrollment
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control Group | Weight Loss Group
Number analyzed (Participants) | 0 | 5
ng/ml
  Baseline Leptin |  | 39.5 (7.7)
  Week 8 Leptin |  | 13.4 (1.6)

2. Primary Outcome: The Primary Outcome Will be Insulin Levels at Baseline and 8 Weeks
Description: The secondary outcome was deleted, since it was finally not performed in the study due to problems in enrollment
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: μU/ml
Arm/Group | Control Group | Weight Loss Group
Number analyzed (Participants) | 0 | 5
μU/ml
  Baseline Insulin |  | 13 (1.6)
  Week 8 Insulin |  | 6.4 (1.4)

3. Primary Outcome: The Primary Outcome Will be HOMA-IR at Baseline and 8 Weeks
Description: The secondary outcome was deleted, since it was finally not performed in the study due to problems in enrollment
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: HOMA score
Arm/Group | Control Group | Weight Loss Group
Number analyzed (Participants) | 0 | 5
HOMA score
  Baseline HOMA-IR |  | 2.82 (0.37)
  Week 8 HOMA-IR |  | 1.33 (0.31)

ADVERSE EVENTS:
Arm/Group | Control Group | Weight Loss Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/5
Other Adverse Events (participants affected / at risk) | 0/0 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No